CLINICAL TRIAL: NCT07393334
Title: Effects of NLS-133, a Potential Non-Hormonal "On-Demand" Male Contraceptive, on Semen Volume and Sperm Count in Normal Men: A Double-Blind, Placebo-Controlled Trial
Brief Title: Effects of NLS-133, a Potential Non-Hormonal "On-Demand" Male Contraceptive
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Next Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLS-133-CLIN001
Record Dates: First submitted 2025-12-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Male Contraception; Semen Volume; Sperm Motility
Keywords: Effect of NLS-133 on semen volume and semen parameters

STUDY DESIGN:
Intervention Model Description: Randomized, placebo- and active-controlled, cross-over design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Active Control (Active Comparator): generic alpha-1-adrenergic receptor antagonist
  Interventions: Drug: Active Comparator #1
- NLS-133 (combination of two FDA-approved drugs) (Experimental)
  Interventions: Drug: NLS-133

INTERVENTIONS:
Drug: NLS-133 — NLS-133 is the primary experimental arm of the study
  Arms: NLS-133 (combination of two FDA-approved drugs)
Drug: Placebo — Double placebo arm of the study
  Arms: Placebo
Drug: Active Comparator #1 — Active control arm of study
  Other Names: Active control
  Arms: Active Control

SUMMARY:
NLS-133-CLIN001 is a Phase 2a study designed to assess the safety, tolerability, and effects of NLS-133 (combination of two FDA-approved agents) compared to an active control (FDA-approved pharmacologic agent) or placebo on semen volume and sperm count in 10 in healthy men. Participants will be randomized in a crossover design to receive a single dose of NLS-133, an active control or placebo either 90 or 180 minutes prior to collection of semen. Sperm parameters measured will be count, motility and morphology. A brief questionnaire will be completed by each subject during each treatment cycle that addresses orgasm and ejaculation quality. Safety monitoring will include adverse event reporting, laboratory assessments, and vital signs.

DETAILED DESCRIPTION:
The aim of study NLS-133-CLIN001is to determine the time frame NLS-133 (combination of two FDA-approved agents) affected ejaculation, semen volume and sperm count in young, normal men. NLS-133 responses will be compared to responses observed after oral placebo and active control (FDA-approved pharmacological agent) treatments. This is a randomized, double-blind, placebo-controlled, crossover (6-way) trial of 10 men who will receive oral capsules 90 and 180 minutes prior to semen collection by masturbation. There will be at least a 72 hour washout period between dosing cycles. Semen volume, if any, and sperm count and morphology (if possible based on semen volume) will be assessed. Subjects will also answer a brief questionnaire regarding orgasm and ejaculation quality during masturbation. Lastly, time to ejaculation and orgasm will be measured by a stopwatch to determine any impact on the time to orgasm or ejaculation by the study treatments. A brief questionnaire about orgasm and ejaculation quality will be completed subjects during each treatment cycle. Safety monitoring will include adverse event reporting, laboratory assessments, and vital signs.

Statistical analyses will be as follows. Means and standard deviations will be calculated for ejaculate volumes and sperm counts at each time point after dosing, stratified by dose. The main outcome for this study is the Semen volume and total sperm count by dose at each time point. This outcome will be compared by Friedman's ANOVA with a Dunnett's post-hoc test. Secondary outcomes include time to ejaculation by dose and orgasm quality scores using the Derogatis questionnaire and other questions as well as serum silodosin and guanfacine concentrations by dose and time and will also be analyzed by Friedman's ANOVA with a Dunnett's post-hoc test. All analyses will be performed using STATA version 10, (College Park, TX). For all comparisons an alpha of <0.05 without correction for multiple comparisons will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age 18-55.
2. Normal physical examination and testicular volume >15 cc
3. No significant medical history that would impact the safety of the study.
4. No current use of drugs that comprise NLS-133
5. Normal values on baseline hematology, blood chemistry and liver function tests and serum testosterone.
6. Normal baseline sperm parameters (semen volume >1.4 cc, sperm concentration >15 million/ml, motility >40% and morphology >4%).
7. Willing and able to comply with all study requirements and procedures.

Exclusion Criteria:

1. History or evidence of erectile dysfunction.
2. Inability to produce semen samples in clinic setting.
3. Significant chronic or acute medical illness.
4. Previous or current ethanol or illicit drug abuse.
5. Evidence of significant underlying disease (based on results of the physical exam and the routine labs).
6. Known infertility or hypogonadism.
7. Planned or anticipated use of any prohibited medications during participation in the study. These include use of sex hormones for treatment, testosterone, anabolic steroids, retinoic acid (e.g., Accutane®), vitamin A, other drugs known to inhibit spermatogenesis, opioids, cocaine, methamphetamine, and/or the consumption of >4 alcoholic beverages daily.
8. Presence of moderate-to-severe pulmonary or cardiovascular disease
9. Known active hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or COVID-19 infection.
10. History of malignancy within 5 years before the Screening Visit, except fully treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
11. Known active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antifungals, antiparasitics or antiprotozoals during the Screening period.
12. Any other acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with study participation in the judgment of the investigator would make the participant inappropriate for entry into the study.
13. Participation in another investigational clinical trial within the last 30 days.
14. Participants who live in detention on court order or on regulatory action.
15. Related to sponsor or staff involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Semen volume (mL) | 90 and 180 minutes for each treatment cycle
Sperm count (millions/mL) | 90 and 180 minutes for each treatment cycle
  Measurement of sperm count

SECONDARY OUTCOMES:
Sperm motility | 90 and 180 after placebo, active-control or NLS-133 administration
  Total percentage of sperm that are actively swimming

CONTACTS AND LOCATIONS:
Locations (1):
- Population Center for Research in Human Reproduction and Departments of Medicine, University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Small-scale (10 subjects) proof of concept study